CLINICAL TRIAL: NCT06985134
Title: Comparative Efficacy and Safety of Thalidomide and Sulfasalazine in Moderate to Severe Ankylosing Spondylitis: A Real-World Study From Bangladesh
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, A F M Mahbubul Alam, Assistant professor, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1638
Record Dates: First submitted 2025-05-13; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2017-01

CONDITIONS: Comparative Efficacy and Safety of Thalidomide and Sulfasalazine in Moderate to Severe Ankylosing Spondylitis: A Real-World Study From Bangladesh; Condition ...Moderate to Severe Axial Spondyloarthopathy
MeSH Terms: interventions — Sulfasalazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comparative Efficacy and Safety of Thalidomide and Sulfasalazine in Moderate to Severe Ankylosing Sp (Experimental)
  Interventions: Drug: Comparative Efficacy and Safety of Thalidomide and Sulfasalazine in Moderate to Severe Ankylosing Spondylitis: A Real-World Study from Bangladesh

INTERVENTIONS:
Drug: Comparative Efficacy and Safety of Thalidomide and Sulfasalazine in Moderate to Severe Ankylosing Spondylitis: A Real-World Study from Bangladesh — The present study included patients aged >18 years with inflammatory low back pain fulfilling the Modified New York criteria [12], 2014 for moderate to severe ankylosing spondylitis. The criteria include radiographic sacroiliitis (at least grade II bilaterally or grade III unilaterally) along with clinical signs, such as inflammatory back pain for at least 3 months' duration, limitation of lumbar spine in sagittal and frontal planes, or chest expansion decreased relative to normal values for age and sex. Exclusion criteria were non-inflammatory back pain or back pain due to inflammatory causes other than AS, failure to confirm a washout period of four weeks, those who were on DMARDs, allergy to thalidomide, Sulfasalazine, and NSAIDs, known to have kidney diseases or cardiac disease, active peptic ulcer disease, and pregnancy.

SUMMARY:
the present study was conducted to determine the comparative efficacy and safety of thalidomide and SSZ in moderate to severe cases of ankylosing spondylitis in Bangladesh.

ELIGIBILITY:
Inclusion Criteria:

* The present study included patients aged >18 years with inflammatory low back pain fulfilling the Modified New York criteria for moderate to severe ankylosing spondylitis. The criteria include radiographic sacroiliitis (at least grade II bilaterally or grade III unilaterally) along with clinical signs, such as inflammatory back pain for at least 3 months' duration, limitation of lumbar spine in sagittal and frontal planes, or chest expansion decreased relative to normal values for age and sex

Exclusion Criteria:

* Exclusion criteria were non-inflammatory back pain or back pain due to inflammatory causes other than AS, failure to confirm a washout period of four weeks, those, those who were on DMARDs, allergy to thalidomide, sulphasalazine, and NSAIDs, known to have kidney diseases or cardiac disease, active peptic ulcer disease, and pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
BASDAI | Outcome 1: "Bath Ankylosing Spondylitis Disease Activity index(BASDAI) pain score at baseline"; Outcome 2: " "Bath Ankylosing Spondylitis Disease Activity index(BASDAI) pain score at week 12""
  score of this scale is o to 10. o means no pain and 10 means maximum pain

CONTACTS AND LOCATIONS:
Overall Officials: ISLAM, Study Director — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Bsmmu, Dhaka, Shahbag, Bangladesh

IPD SHARING:
Plan to Share IPD: No